CLINICAL TRIAL: NCT00000724
Title: A Study of Trimetrexate With Leucovorin Rescue for AIDS Patients Who Are Refractory to Standard Therapies for Pneumocystis Carinii Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NS 401
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimetrexate; Pneumonia, Pneumocystis carinii; Injections, Intravenous; Leucovorin; Drug Evaluation; Drug Therapy, Combination; Folic Acid Antagonists; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Leucovorin calcium

SUMMARY:
To study the safety and effectiveness of trimetrexate (TMTX) plus leucovorin calcium rescue (LCV) in the treatment of Pneumocystis carinii pneumonia (PCP) in patients who have AIDS, patients who are HIV positive, or those for whom laboratory confirmation of HIV infection has not yet been established if they are at high risk for HIV infection, and who have not responded to standard treatments or who have demonstrated severe or life-threatening intolerance to both conventional therapies for PCP.

The drugs trimethoprim / sulfamethoxazole (TMP / SMX) and pentamidine, usually used to treat PCP in AIDS patients, have proven ineffective in many patients and have had to be discontinued in many other patients because of severe side effects. TMTX was chosen for this trial because it was found to be very active against the PCP organism in laboratory tests and, in a preliminary trial in combination with LCV, there was a high response rate without severe toxicity.

DETAILED DESCRIPTION:
The drugs trimethoprim / sulfamethoxazole (TMP / SMX) and pentamidine, usually used to treat PCP in AIDS patients, have proven ineffective in many patients and have had to be discontinued in many other patients because of severe side effects. TMTX was chosen for this trial because it was found to be very active against the PCP organism in laboratory tests and, in a preliminary trial in combination with LCV, there was a high response rate without severe toxicity.

AMENDED: 08/01/90. As of August 31, 1989, 437 patients were enrolled into uncontrolled studies of trimetrexate for PCP: 214 in TX 301/ACTG 039 (trimetrexate for patients intolerant of approved therapies) and 223 in NS 401 (trimetrexate for patients refractory to approved therapies). The analysis of overall response rate, stringently defined as having received at least 14 days of trimetrexate and being alive at follow-up 1 month after the completion of therapy, reveals 84/159 intolerant patients and 48/160 refractory patients had responded, for rates of 53 percent and 30 percent, respectively. These response rates include all individuals who received at least one dose of trimetrexate. Of the 111 patients who were ventilator-dependent at study entry, 18 completed a course of therapy and were alive a month later, for a response rate of 16 percent. All other ventilated patients died. The most common severe (grades 3 and 4) toxicities were: transaminase elevation (> 5 x normal) in 94 patients, anemia (< 7.9 g/dl) in 109, neutropenia (< 750 cells/mm3) in 58, fever (> 40 C) in 37, and thrombocytopenia (< 50000 platelets/mm3) in 27.

Toxicity required discontinuation of therapy in approximately 5 percent of all patients. Original design: Patients entered in the study are given TMTX once a day for 21 days and LCV 4 times a day (every 6 hours) for 24 days. Doses are determined by body size. Both drugs are given by intravenous infusion, but LCV may be given orally after the first 10 days. Doses are adjusted if side effects, such as low white blood cell count, are too severe. During the 21-day trial, zidovudine (AZT) may not be used, because of possible increased bone marrow toxicity. AZT may be resumed as soon as the administration of TMTX and LCV has been completed. After treatment with TMTX, the patient may be treated with other drugs to prevent the recurrence of PCP at the discretion of his/her physician.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antihypertensive agents.

Concurrent Treatment:

Allowed:

* Blood products.
* Ventilatory support.

Prior Medication:

Required:

* At least 7 days trimethoprim / sulfamethoxazole or parenteral pentamidine.
* Allowed:
* Myelosuppressive or nephrotoxic agents including zidovudine, but must be discontinued during trial.

No improvement in ventilatory status, defined as no change or a decrease in arterial or alveolar difference ((A-a) DO2) in the 72 hours prior to entry. (A-a) DO2 should be determined on room air, or receiving an FiO2 of 100 percent for 10 minutes via a tightly fitting non-rebreathing mask, or at an FiO2 of 100 percent for 10 minutes if the patient is being ventilated. Intolerance to TMP / SMX is defined as one or more of the following:

* Platelets < 50000 platelets/mm3 or absolute neutrophil count (polys + bands) = or < 500 cells/mm3 on at least two occasions = or > 12 hours apart.
* Blistering rash, mucosal involvement, generalized maculopapular eruption or intolerable pruritus.
* Transaminase > 5 x ULN or = or > 300 IU if baseline abnormal.
* Daily temperature = or > 103 degrees F beginning after the 5th day of treatment and persisting for at least 3 days and not responsive to antipyretic therapy, with no other discernible cause.
* Any other severe or life-threatening adverse reaction to TMP / SMX that, in the investigator's opinion, makes continued or recurrent treatment with TMP / SMX inadvisable (approved on a case-by-case basis by the NIAID clinical monitor).
* Intolerance to pentamidine is defined as one or more of the following:
* Platelets < 50000 platelets/mm3 or absolute neutrophil count (polys + bands) < 550 cells/mm3 on at least two occasions = or > 12 hours apart.
* Serum creatinine > 3.0 mg/dl.
* Systolic blood pressure < 90 mm requiring supportive therapy.
* Symptomatic hypoglycemia with blood glucose = or < 40 or hyperglycemia requiring therapy.
* Pancreatitis with laboratory confirmation (abnormal amylase and/or lipase).
* Any other severe or life-threatening adverse reaction to pentamidine that, in the investigator's opinion, makes continued or recurrent treatment with pentamidine inadvisable (approved on a case-by-case basis by the NIAID clinical monitor).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reactions due to trimetrexate.
* Patients with less severe adverse reactions may be enrolled if, in the opinion of the investigator, they do not prohibit rechallenge with the drug.

Concurrent Medication:

Excluded:

* Myelosuppressive or nephrotoxic agents.
* Other investigational drugs including high-dose steroids (exceeding physiologic replacement doses).

Patients with the following are excluded:

* History of Type I hypersensitivity (i.e., urticaria, angioedema, or anaphylaxis), exfoliative dermatitis, or other life-threatening reactions due to trimetrexate.
* Patients with less severe adverse reactions may be enrolled if, in the opinion of the investigator, they do not prohibit rechallenge with the drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (1):
- Warner-Lambert Parke-Davis, Morris Plains, New Jersey, United States

REFERENCES:
- [Background] Feinberg J, McDermott C, Nutter J. Trimetrexate (TMTX) salvage therapy for PCP in AIDS patients with limited therapeutic options. Int Conf AIDS. 1992 Jul 19-24;8(2):B136 (abstract no PoB 3297)